CLINICAL TRIAL: NCT00005120
Title: A Phase IB Study to Evaluate the Safety, Pharmacokinetics, and Effects of (+)-Calanolide A on Surrogate Markers in HIV-Positive Patients With No Previous Antiretroviral Therapy
Brief Title: The Safety and Effectiveness of (+)-Calanolide A in HIV-Infected Patients Who Have Never Taken Anti-HIV Drugs
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sarawak MediChem Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 297B; 57CL-0001
Record Dates: First submitted 2000-04-20; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-06

CONDITIONS: HIV Infections
Keywords: CD4 Lymphocyte Count; Biological Markers; Anti-HIV Agents; Viral Load; Pharmacokinetics; calanolide A
MeSH Terms: conditions — HIV Infections | interventions — calanolide A

INTERVENTIONS:
Drug: Calanolide A

SUMMARY:
The purpose of this study is to see if it is safe and effective to give calanolide A to HIV-infected adults who have not used anti-HIV drugs in the past.

DETAILED DESCRIPTION:
Patients are randomized to receive (+)-calanolide A or placebo for 21 days. All patients may elect to receive an open-label, 3-month course of approved retroviral therapy (up to triple-drug therapy) to be selected by, and administered under the care of, the patients' physicians. If the patient has no insurance coverage or does not wish to utilize his/her insurance for anti-HIV medications, Sarawak MediChem Pharmaceuticals will provide these medications at no charge for up to 3 months.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 18 years old.
* Agree to use effective methods of birth control during the study.
* Have a CD4 cell count of 200 cells/mm3 or more.
* Have HIV levels of 5000 copies/ml or more.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have abnormal blood tests.
* Have had a reaction to study medication.
* Have a history of opportunistic (AIDS-related) infection or cancer.
* Are being treated for active pulmonary tuberculosis.
* Have a fever of 39 degrees C or more within 14 days of beginning study treatment.
* Are unable to take medications by mouth.
* Have an abnormal chest X-ray or ECG within 30 days of beginning study treatment.
* Have hepatitis, hemophilia, or other blood disorder.
* Have significant heart, stomach, intestinal, liver, nerve, or kidney problems.
* Have a condition which may affect ability to participate in this study, such as drug or alcohol abuse or a serious mental disorder.
* Have taken anti-HIV drugs in the past.
* Are taking certain medications.
* Have had a blood transfusion within the 3 months prior to entering the study.
* Have had radiation or chemotherapy within 16 days before the screening visit or plan to receive such treatment during the study.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2000-04

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - South Florida Bioavailability Clinic, Miami, Florida
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Anderson Clinical Research, Philadelphia, Pennsylvania
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Burnside Clinic, Columbia, South Carolina
  - Univ of Texas Med Branch, Galveston, Texas